CLINICAL TRIAL: NCT05457764
Title: Does Erotica by Virtual Reality Improve Sperm Quality
Brief Title: Erotica by Virtual Reality on Sperm Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryos International (Industry)
Responsible Party: Principal Investigator, Daniel Rosenkjær, Research Scientist, Cryos International
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VRStudy
Record Dates: First submitted 2022-06-27; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Virtual Reality
Keywords: ejaculate quality; virtual reality; male fertility; sperm donation; erotic stimulation

STUDY DESIGN:
Intervention Model Description: Balanced and randomized controlled cross-over within-subjects design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants use Virtual reality headsets as medium of erotica to produce their sperm sample
  Interventions: Device: Virtual reality headset
- No Virtual Reality (No Intervention): Participants did not use Virtual reality headsets as medium of erotica to produce their sperm sample. They used a computer screen to display erotica.

INTERVENTIONS:
Device: Virtual reality headset — The VR headset was a Pico G2, Pico Interactive, San Fransisco, USA, offering a choice from 60 erotic videos each of 10-30 minutes duration. The men were allowed to watch any and as many of these video clips as they wished. The "No VR" arm, donors used the computer monitor available in the donation rooms.
  Arms: Virtual Reality

SUMMARY:
Objective To study whether erotica by virtual reality (VR) during masturbation influences the quality of sperm donor ejaculates.

Hypothesis Erotica by virtual reality improves ejaculate quality.

DETAILED DESCRIPTION:
The study design was within-subjects repeated measures, using balanced, randomized, controlled, cross-over sampling. Data was collected between 1 August and 25 November 2021 in the four largest cities in Denmark (Copenhagen, Aarhus, Odense, and Aalborg) from consenting sperm donors at Cryos International. A total of 63 'accepted' donors (aged 19 - 44 years old and with a BMI between 17 to 35) participated in the study.

The VR setup involved a headset (Pico G2, Pico Interactive, San Fransisco, USA) offering a choice from 60 erotic videos each of 10-30 minutes duration. The men were allowed to watch any and as many of these video clips as they wished.

Sperm samples were donated in private rooms dedicated for the purpose and equipped with a touch screen showing erotic material. The men were asked to donate as usual and self-report the amount of time (in hours) since their last ejaculation (the abstinence period). Every other donation, donors rolled dice to determine whether a VR headset would be used; with the subsequent donation performed with the opposite condition. To maximize privacy and minimize stress on the donors, the amount of time the donors took to produce a sperm sample (donation period) was recorded as the number of seconds from closing the door to the private room to when it was opened again.

Each semen sample was weighed to determine ejaculate volume and allowed to liquify at room temperature for up to 1 hour. After liquefaction, aliquots were loaded in duplicate onto Makler counting chambers (Sefi-Medical, Israel) and observed at 200x magnification using an Olympus CX41 microscope (Olympus, Japan). Measurements of sperm concentration, motility and motile sperm concentration were made using a MICROPTIC, S.L. (Barcelona, Spain) Computer Assisted Sperm Analysis system with at least 500 cells counted per analysis. No analysis of sperm morphology was performed.

The investigators used linear mixed models (LMMs) to assess the relationship between VR-use and ejaculate volume, donation period and total motile sperm count (TMSC) for each ejaculate sample, while controlling for several factors that might also influence ejaculates: (i) abstinence period, (ii) donor age, (iii) donor BMI, (iv) day of the year (season), and (v) location (donation site). In each model, the investigators included anonymized donor identity as a random effect to avoid pseudo-replication as each donor provided multiple samples. The interaction between VR-use and abstinence period was initially included in models as abstinence period is known to increase ejaculate size and quality, though sometimes a decrease has been observed. The investigators considered it to be at least plausible that the influence of VR might diminish as abstinence period increased and both ejaculate size and quality approached their maxima for each donor. The investigators removed those interaction terms from models when p-values for the interactions was >0.20.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to donate at least 3 samples for each study arm (i.e. minimum 6 samples total).
* Must be an 'accepted' donor at Cryos International i.e. must have a post thaw sperm concentration of ≥5x106 per ml.

Exclusion Criteria:

* Not an 'accepted' donor at Cryos International

Ages: 19 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Total motile sperm count | Within 1 hour of ejaculate sample procurement
  The total number of motile sperm cells in the ejaculate. Counted by computer assisted sperm analyzer

SECONDARY OUTCOMES:
Donation time | Within 120 minutes of commencement of donation of sample
  The time of which the sperm donors used in the donation rooms to produce the sperm sample

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rosenkjær, Principal Investigator — Research Scientist
Locations (4):
- Denmark (4):
  - Cryos International - Aalborg ApS, Aalborg
  - Cryos International - Aarhus ApS, Aarhus C
  - Cryos International - København ApS, Copenhagen
  - Cryos International - Odense ApS, Odense

IPD SHARING:
Plan to Share IPD: No
The data will be publicly available on figshare.com, but in anonymized form so that IPD cannot be discerned.

REFERENCES:
- [Derived] Rosenkjaer D, Pacey A, Montgomerie R, Skytte AB. Effects of virtual reality erotica on ejaculate quality of sperm donors: a balanced and randomized controlled cross-over within-subjects trial. Reprod Biol Endocrinol. 2022 Oct 11;20(1):149. doi: 10.1186/s12958-022-01021-1. PMID 36221120

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT05457764/Prot_SAP_000.pdf